CLINICAL TRIAL: NCT03134027
Title: Reconstitution of a Human Immune System in a Patient Derived Xenograft (PDX) Model of Genitourinary (GU) Cancers
Acronym: Immune PDX
Status: Terminated | Type: Observational
Why Stopped: Poor accrual
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00082398
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Genito Urinary Cancer; Bladder Cancer; Kidney Cancer; Prostate Cancer
MeSH Terms: conditions — Urogenital Neoplasms; Urinary Bladder Neoplasms; Kidney Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects from which PDXs have been generated.: Subjects will be identified from which PDXs have been generated from an already approved IRB protocol.
  Interventions: Procedure: Bone marrow biopsy
- Subjects without an existing PDX: Subjects with prostate cancer amenable to a tumor biopsy.
  Interventions: Procedure: Tumor biopsy

INTERVENTIONS:
Procedure: Bone marrow biopsy — Subjects will undergo a bone marrow biopsy to obtain aspirate for stem cell collection.
  Groups: Subjects from which PDXs have been generated.
Procedure: Tumor biopsy — Subjects will undergo a tumor biopsy to obtain tissue for generation of a PDX.
  Groups: Subjects without an existing PDX

SUMMARY:
The objective of this study is to obtain human blood CD34+ hematopoietic stem/progenitor cells (HSPCs) to reconstitute a match human immune system in our PDX model. The hypothesis is that by using matched leukocytes and PDX from the same patient, rejection of the PDX by the host immune system will not be observed and therefore a preclinical model to study immunotherapy can be developed to study, understand and improve upon our current therapies. HSPCs will be collected from bone marrow aspirate obtained from a bone marrow biopsy.

The secondary objective is to use patient tumor biopsy samples or circulating tumor cell samples to develop additional preclinical models of GU cancers, particularly prostate cancer, that are clinically relevant by generating additional PDXs.

ELIGIBILITY:
Inclusion Criteria for Bone Marrow Biopsy:

1. Patients with Genitourinary (GU) Cancers and presence of existing patient derived xenograft or planned collection of tumor for PDX generation
2. Age ≥ 18 years.
3. Ability to understand and provide signed informed consent that fulfills Institutional Review Board guidelines.
4. Ability to undergo bone marrow biopsy
5. Laboratory requirements (Hematocrit 30%, Platelets 75,000 + 10^6/l and WBC 4000 X 10^6/l)
6. Karnofsky performance status >70%

Exclusion Criteria for Bone Marrow Biopsy:

1. Participants with serious concurrent chronic or acute illness that would affect the safety of a bone marrow biopsy.

Inclusion Criteria for Tumor Biopsy

1. Patients with prostate cancer

   a. Biopsies in this study for diseases other than prostate cancer are not permitted.
2. Age ≥ 18 years.
3. Ability to understand and provide signed informed consent that fulfills Institutional Review Board guidelines.
4. Planned or willing to undergo a tumor biopsy. Biopsies may be for research or clinical purposes depending on the treating provider for men with prostate cancer. Biopsies in this study for diseases other than prostate cancer are not permitted

   1. For research only biopsies: At least one lymph node or bone metastatic amenable to a minimum risk biopsy in the opinion of the treating physician.
   2. For clinical purpose biopsies: There are no location or risk requirements.
5. Laboratory requirements (Hematocrit 30%, Platelets 75,000 X 10^6/l and WBC 4000 X 10^6/l)
6. Karnofsky performance status >70%

Exclusion Criteria for Tumor Biopsy:

1. Participants with serious concurrent chronic or acute illness that would affect the safety of a tumor biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Duke Cancer Institute Patients
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
Reconstitution of a matched human immune system in patient derived xenografts (PDXs) | approximately 4 months
  Number of samples yielding a matched human immune system in immunodeficient mice resulting in a PDX with a humanized immune system.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Armstrong, MD, ScM, Principal Investigator — Duke Cancer Institute
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States